CLINICAL TRIAL: NCT03457233
Title: The Impact of Overweight and Obesity on Reproductive Outcomes in Poor Ovarian Responders in ICSI Cycles
Brief Title: The Impact of Body Weight on Reproductive Outcomes in Poor Ovarian Responders in ICSI Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 31
Record Dates: First submitted 2018-02-25; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Invitro Fertilization
MeSH Terms: interventions — Gonadotropins; Menotropins; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal weight (Active Comparator): 18.5- 24.9 kg/m2
  Interventions: Drug: Gonadotropins; Drug: GNRH antagonist; Drug: Human chorionic gonadotropin Chorimon; Drug: Natural progesterone
- Overweight (Active Comparator): BMI 25-29.9 kg/m2
  Interventions: Drug: Gonadotropins; Drug: GNRH antagonist; Drug: Human chorionic gonadotropin Chorimon; Drug: Natural progesterone
- Obese (Active Comparator): BMI ≥ 30 kg/m2
  Interventions: Drug: Gonadotropins; Drug: GNRH antagonist; Drug: Human chorionic gonadotropin Chorimon; Drug: Natural progesterone

INTERVENTIONS:
Drug: Gonadotropins — 1) Gonadotrophines is started on day 2 with HMG(merional, IBSA) ,until the day of HCG administration
  Other Names: Human menopausal gonadotropin
Drug: GNRH antagonist — cetrorelix 0,25mg s.c is given using flexible protocol, it is given when at least one follicle reaches size 14 mm to prevent premature lutenization ,until the day of hCG administration
  Other Names: cetrorelix
Drug: Human chorionic gonadotropin Chorimon — 10000 IU of HCG are given intramuscular when 2 or more mature follicles reach 18 - 20 mm
  Other Names: HCG
Drug: Natural progesterone — 400 mg vaginal tablets twice daily from the day of ovum pick up till HCG tesing
  Other Names: prontogest

SUMMARY:
Induction of ovulation cycle:

1. Gonadotrophines is started on day 2 with HMG(merional, IBSA) ,until the day of HCG administration(choriomon,IBSA10000IU) with starting dose 300 to 450iu.
2. GNRH antagonist (cetrorelix 0,25mg s.c, cetrotide, serono laboratories, Aubonne Switzerland) is given using flexible protocol, it is given when at least one follicle reaches size 14 mm to prevent premature lutenization ,until the day of hCG administration
3. Ovarian ultrasound scans were performed using a 5.0-9.0 MHZ multi frequency trans vaginal probe (mindrayDP-5)to assess the ovarian response till the mature follicles reach18-20mm when hCG administration 10000 IU is given.Serum E2 level is done on day of HCG trigger.
4. Trans vaginal ultrasound-guided oocyte retrieval is performed 34-36 hours after hCG injection
5. Progesterone vaginal tablets (Prontogest,IBSA) are administrated 400mg twice daily as luteal support from the day of oocytes retrieval.
6. Ultrasound -guided fresh embryo transfer is performed on day 2 or 3 after fertilization.
7. Serum hCG assessment to detect pregnancy is performed at 14 days after embryo transfer .if positive(chemical pregnancy) ,women undergo trans -vaginal ultrasonography 2 weeks after, to confirm fetal pulsations as well as number of gestational sacs (clinical pregnancy).
8. The implantation rate is calculated as the number of viable embryos divided by the number of transferred embryos multiplied by 100

DETAILED DESCRIPTION:
Induction of ovulation cycle:

1. Gonadotrophines is started on day 2 with HMG(merional, IBSA) ,until the day of HCG administration(choriomon,IBSA10000IU) with starting dose 300 to 450iu.
2. GNRH antagonist (cetrorelix 0,25mg s.c, cetrotide, serono laboratories, Aubonne Switzerland) is given using flexible protocol, it is given when at least one follicle reaches size 14 mm to prevent premature lutenization ,until the day of hCG administration
3. Ovarian ultrasound scans were performed using a 5.0-9.0 MHZ multi frequency trans vaginal probe (mindrayDP-5)to assess the ovarian response till the mature follicles reach18-20mm when hCG administration 10000 IU is given.Serum E2 level is done on day of HCG trigger.
4. Trans vaginal ultrasound-guided oocyte retrieval is performed 34-36 hours after hCG injection
5. Progesterone vaginal tablets (Prontogest,IBSA) are administrated 400mg twice daily as luteal support from the day of oocytes retrieval.
6. Ultrasound -guided fresh embryo transfer is performed on day 2 or 3 after fertilization.
7. Serum hCG assessment to detect pregnancy is performed at 14 days after embryo transfer .if positive(chemical pregnancy) ,women undergo trans -vaginal ultrasonography 2 weeks after, to confirm fetal pulsations as well as number of gestational sacs (clinical pregnancy).
8. The implantation rate is calculated as the number of viable embryos divided by the number of transferred embryos multiplied by 100

ELIGIBILITY:
Inclusion Criteria:

* 4- Poor responder according to ESHRE consensus; in which at least 2 of the following should be present: Advanced maternal age (≥ 40 years old) or any other risk factor A previous poor ovarian response (cycles cancelled or ≤ 3 oocytes with a conventional protocol)An abnormal ovarian reserve test (ORT); antral follicle count (AFC) < 5-7 follicles or anti-mullerian hormone (AMH) ≤0.5- 1.1 ng/ml In the absence of advanced maternal age or abnormal ORT, two previous episodes of poor ovarian response after maximal stimulation patients are also considered poor responders according to ESHRE consensus.

Presence and Adequate visualization of both ovaries Uterine cavity within normal anatomy assessed with HSG, hysteroscopy and TVUS

Exclusion Criteria:

Any factor which may affect reproductive outcome other than that the patient is a poor responder will be excluded from the study, like:

1. Severe male factor .
2. Uterine factor (eg: fibroid, polyp, Ashermann, .. etc)
3. Immunological disorder (eg: SLE, APS, … etc)
4. Thyroid or adrenal dysfunction
5. Neoplasia (especially: hypothalamic, pit, ovarian)
6. Women diagnosed with PCOS according to Rotterdam criteria
7. Hydrosalpinx that hasn't been surgically removed or ligated.
8. Untreated hyperprolactinemia
9. Abnormal bleeding disorder
10. Hepatic or renal dysfunction
11. Hypersenstivity to study medication ( GNRH antagonist)
12. Need to take medication that can influence ovarian stimulation
13. Endometriosis grade 3 or 4
14. Ovarian cyst> 10 cm.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 185 (Estimated)
Dates: Start 2015-01-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks after HCG triggering
  appearance of intrauterine gestational sac by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Fahmy RM, Rashwan H, Mahmood M, Hassan SM, Nabil H, Hany A, Lotfy R, Lasheen YS, Dahab S, Darwish M. Effect of body mass index on the outcome of IVF cycles among patients with poor ovarian response. Int J Gynaecol Obstet. 2019 Feb;144(2):161-166. doi: 10.1002/ijgo.12706. Epub 2018 Nov 26. PMID 30407618